CLINICAL TRIAL: NCT04186312
Title: Improving the Educational and Social-Emotional Functioning of College Students With ADHD
Brief Title: A Psychosocial Treatment Program for College Students (ACCESS)
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arthur Anastopoulos, Principal Investigator, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 15-0216
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial comparing Immediate versus Delayed Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Cognitive-Behavioral Treatment program known as ACCESS
  Interventions: Behavioral: ACCESS - Accessing Campus Connections & Empowering Student Success
- Delayed Treatment (Other): Allowed to receive treatment as usual during study, then received ACCESS after delay of two-semesters
  Interventions: Behavioral: ACCESS - Accessing Campus Connections & Empowering Student Success

INTERVENTIONS:
Behavioral: ACCESS - Accessing Campus Connections & Empowering Student Success — Cognitive-Behavioral Treatment delivered across 2 semesters via group and individual mentoring sessions

SUMMARY:
The results of this study are expected to provide important and new information regarding the treatment of academic impairment among college students with ADHD. The present study should provide a substantial addition to the existing knowledge base concerning interventions for college students with ADHD. In addition, because the intervention is being implemented during college, potential benefits include the prevention of the severe academic and psychosocial functioning difficulties associated with ADHD, including school dropout.

DETAILED DESCRIPTION:
This proposal, "Improving the Educational and Social-Emotional Functioning of College Students with ADHD," was submitted in response to CFDA-84.305A Postsecondary and Adult Education Research, Goal 3 - Efficacy and Replication.

The number of young adults with Attention-Deficit/Hyperactivity Disorder (ADHD) pursuing college degrees has increased dramatically over the past 30 years. Students with ADHD currently represent one of the largest disability groups on college campuses, with at least 25% of all college students who receive disability services identified with ADHD. The need for such services is clearly warranted, given that college students with ADHD are at increased risk for having low and failing grades, being placed on academic probation, and ultimately dropping out of college. Currently, many colleges and universities offer students with ADHD extended time and other accommodations. Unfortunately, use of these accommodations is not empirically supported, presumably because they do not address the core difficulties - deficits in executive and psychological functioning - shown to lead to educational impairment in college students with ADHD. Further complicating matters is that systematic investigation of potentially useful psychosocial interventions for college students with ADHD has been lacking.

The investigators set out to address this gap by working with stakeholders to develop a psychosocial intervention for college students with ADHD, known as ACCESS - Accessing Campus Connections and Empowering Student Success. Development of ACCESS was guided by careful consideration of conceptual and empirical factors thought to contribute to the difficulties experienced by college students with ADHD, thus resulting in an intervention that specifically targets executive functioning, other core ADHD features, and psychological functioning. To date, a detailed treatment manual has been developed and revised through an iterative process. A large open trial of ACCESS was recently completed by one of the PIs and a second open trial of a similar intervention was independently completed by the other PI. These trials demonstrate the feasibility of delivering ACCESS on college campuses with fidelity and establish preliminary efficacy. In both trials, college students with ADHD made significant improvements in ADHD symptom severity, executive functioning, educational performance, and emotional functioning. Although promising, such findings are limited by the absence of control groups, thereby preventing firm conclusions about efficacy. Accordingly, the primary goal of this Goal 3 study is to conduct a multi-site randomized controlled trial to evaluate the efficacy of the ACCESS intervention and to assess moderators and mediators of intervention response.

College students with ADHD (N=240) from two large, diverse public universities were randomly assigned either to ACCESS or to a delayed treatment condition. Five cohorts of students were recruited, with each cohort consisting of 24 students from each site. Educational, executive, psychological, and social functioning, as well as service utilization, were assessed at pre-treatment, at the end of active intervention, at the end of the maintenance phase, and during a 6-month follow-up. An intent-to-treat analysis was used to assess the efficacy of ACCESS. Moderator and mediator analyses will also be conducted to address the types of students most likely to benefit from ACCESS and to evaluate key mechanisms of change that lead to improved academic and social-emotional functioning.

This study has significant potential to improve the performance of college students with ADHD because the intervention was specifically designed to address deficits in executive and psychological functioning, factors shown to predict the educational outcomes of college students with ADHD. Further, the ACCESS intervention was designed with stakeholder input and thus has clear potential for dissemination upon proof of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* voluntary consent
* 18-30 years of age
* DSM-5 criteria for ADHD
* estimated IQ greater than 85

Exclusion Criteria:

* co-occurring autism spectrum disorder, bipolar disorder, obsessive-compulsive disorder, and/or active substance abuse

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Conners' Adult ADHD Rating Scale: DSM-IV Inattention Symptom subscale | 4 months, 8 months, 14 months
  Used to assess changes in inattention symptoms, scores range from 0-27, higher scores reflect worse functioning.
Conners' Adult ADHD Rating Scale: DSM-IV Hyperactive-Impulsive Symptom subscale | 4 months, 8 months, 14 months
  Used to assess changes in hyperactive-impulsive symptoms, scores range from 0-27, higher scores reflect worse functioning.
Behavior Rating Inventory of Executive Function, Adult Version - Global Executive Composite subscale | 4 months, 8 months, 14 months
  Used to assess changes in self-reported overall executive functioning, scores range from 70-210, higher scores indicate worse functioning

SECONDARY OUTCOMES:
ADHD Impact Module - Adult: Performance and Daily Functioning subscale | 4 months, 8 months, 14 months
  Used to assess changes in performance and daily functioning, scores range from 0-100, higher scores reflect better functioning.
ADHD Impact Module - Adult: General Well-Being subscale | 4 months, 8 months, 14 months
  Used to assess changes in general well-being, scores range from 0-100, higher scores reflect better functioning.
Learning & Study Strategies Inventory: Test Strategies subscale | 4 months, 8 months, 14 months
  Used to assess self-reported changes in academic functioning, scores range from 8-40, higher scores reflect better functioning.
Learning & Study Strategies Inventory: Study Aids subscale | 4 months, 8 months, 14 months
  Used to assess self-reported changes in academic functioning, scores range from 8-40, higher scores reflect better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur D Anastopoulos, Ph.D., Principal Investigator — UNC Greensboro

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make de-identified data, codebooks, documentation, and research protocols available on UNCG's institutional repository, NC DOCKS (North Carolina Digital Online Collection of Knowledge and Scholarship), through the Odum Institute Data Archive. As an established and trusted repository in the social science field, the Odum Institute Data Archive is a member of the Data Preservation Alliance for the Social Sciences (Data-PASS) and the Library of Congress National Digital Stewardship Alliance (NDSA), and provides a strong archival and data distribution resource to the project. The partnership between NC DOCKS and the Odum Institute allows researchers at UNCG to upload data into the Odum Institute's Dataverse Network at no additional cost to the researcher. Data used for manuscripts accepted and published during or following the grant period will be uploaded and made available at the time the associated manuscripts are first made available by the publisher.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The final, complete data set, including variables that may not have been used in any publications to that point, will be deposited by the project completion date, and made available within 3 years after the end of all data collection activities. All datasets will be stored in, and made available through NC DOCKS for a minimum of 10 years.